CLINICAL TRIAL: NCT07242911
Title: Study on Efficacy and Safety of VMAT Technique With Local Dose Escalation for Unresectable Pancreatic Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Chifeng Tumor Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CFSZLYY-FLK-2025-002
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Ppancreatic Cancer
Keywords: Pancreatic Cancer; VMAT; Radiation Therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dose Escalation Group: Patients with unresectable pancreatic cancer receive Volumetric Modulated Arc Therapy (VMAT) with local dose escalation (total radiotherapy dose 60-65Gy) concurrent with capecitabine chemotherapy.
- Conventional Dose Group: Patients with unresectable pancreatic cancer receive conventional VMAT radiotherapy (total radiotherapy dose 45-50.4Gy) concurrent with capecitabine chemotherapy

SUMMARY:
The goal of this observational study is to learn about the efficacy and safety of the Volumetric Modulated Arc Therapy (VMAT) dose sculpting technique combined with different radiotherapy doses (local dose escalation vs. conventional dose) in patients with unresectable pancreatic cancer, with a focus on survival outcomes, tumor response, and toxic/adverse effects.

The main question it aims to answer is:Does the VMAT dose sculpting technique combined with local dose escalation radiotherapy (total dose 60-65Gy) improve overall survival (OS), progression-free survival (PFS), and tumor response rate while maintaining acceptable safety (i.e., manageable toxic/adverse effects) compared to conventional dose radiotherapy (total dose 45-50.4Gy) in patients with unresectable pancreatic cancer? Participants who have already received VMAT (as part of their regular medical care for unresectable pancreatic cancer) at Chifeng City Cancer Hospital from February 2018 to May 2026 will be divided into two groups based on the radiotherapy dose they received: the study group (local dose escalation, 60-65Gy) and the control group (conventional dose, 45-50.4Gy). All participants will undergo follow-up via phone calls, WeChat, and outpatient re-examinations to collect data on their survival status (OS, PFS), tumor response (assessed by RECIST 1.1 criteria), and toxic/adverse effects (assessed by RTOG for radiation injury and CTCAE 4.0 for chemotherapy-related reactions) until the completion of outcome evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced pancreatic cancer confirmed by pathological diagnosis or PET-CT.
* Patients who refuse surgery or are inoperable.
* No history of radiotherapy.
* Aged 18-76 years with a performance status score of 0-1.

Exclusion Criteria:

* Patients with other concurrent primary malignant tumors.
* Patients unable to tolerate radiotherapy.
* Patients who are unable or unwilling to cooperate with the study.
* Patients with severe dysfunction of vital organs such as liver and kidneys.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: he study population consists of patients with locally advanced pancreatic cancer recruited from Chifeng Tumor Hospital between 2018 and 2026. Inclusion criteria include: pathological or PET-CT confirmed diagnosis, age 18-76 years, Eastern Cooperative Oncology Group (ECOG) performance status 0-1, and no prior radiotherapy. Exclusion criteria are: concurrent other malignant tumors, severe liver/kidney dysfunction, inability to tolerate treatment, and unwillingness to cooperate with the study. Demographic and clinical characteristics such as age, gender, and disease stage will be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in Patients with Unresectable Pancreatic Cancer Treated with VMAT Radiotherapy | Up to 5 years (from February 2018 to May 2026, with follow-up until outcome evaluation completion).
  Time from study enrollment to death from any cause. Assessed via Kaplan-Meier survival analysis using SPSS 27.0, with survival status collected through phone, WeChat, and outpatient follow-up

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) in Patients with Unresectable Pancreatic Cancer Treated with VMAT Radiotherapy | Up to 5 years (from February 2018 to May 2026, with follow-up until outcome evaluation completion).
  Time from study enrollment to tumor progression (per RECIST 1.1 criteria) or death from any cause. Assessed via Kaplan-Meier analysis, with progression status determined by contrast-enhanced CT/MRI every 3 months during follow-up.
Objective Response Rate (ORR) in Patients with Unresectable Pancreatic Cancer Treated with VMAT Radiotherapy | Up to 5 years (from February 2018 to May 2026, with follow-up until outcome evaluation completion).
  Proportion of patients with complete response (CR) or partial response (PR) per RECIST 1.1 criteria. Assessed via contrast-enhanced CT/MRI at 1 month, 3 months, 6 months post-radiotherapy, and every 3 months thereafter, with independent review by two senior radiologists.
Incidence of Chemoradiotherapy Toxicity and Adverse Effects in Patients with Unresectable Pancreatic Cancer Treated with VMAT Radiotherap | Up to 5 years (from February 2018 to May 2026, with follow-up until outcome evaluation completion).
  Incidence of grade ≥2 toxicities/adverse effects related to chemoradiotherapy, assessed by RTOG criteria for radiation injury and CTCAE v4.0 for chemotherapy reactions. Evaluated every 2 weeks during treatment and monthly for 3 months post-treatment, with group comparisons via chi-square test.

CONTACTS AND LOCATIONS:
Locations (1):
- Chifeng Tumor Hospital, Chifeng, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR